CLINICAL TRIAL: NCT07148466
Title: Effects of Scapular and Upper Limb Proprioceptive Neuromuscular Facilitation Techniques on Shoulder Pain, Upper Limb Function & Gait in Stroke With Scapular Dyskinesia.
Brief Title: Scapular and Upper Limb Proprioceptive Neuromuscular Facilitation Techniques in Stroke With Scapular Dyskinesia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aqsa Fayyaz
Record Dates: First submitted 2025-08-24; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Scapular Dyskinesis
Keywords: scapular PNF coupled with upper limb PNF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Experimental): scapular PNF coupled with upper limb PNF and conventional physiotherapy treatment.
  Interventions: Other: Scapular PNF
- GROUP 2 (Active Comparator): Conventional treatment
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Scapular PNF — scapular PNF coupled with upper limb PNF and conventional physiotherapy treatment . It was a 6 week's intervention in which patients got treatment protocol for 30 mints 5 times a week.
  Arms: GROUP 1
Other: Conventional treatment — Conventional treatment. It includes closed kinematic chain exercises of upper limb, upper and lower extremity range of motion exercises, stretching and strengthening exercises for upper limb, trunk and lower limb, balance & coordination, manual dexterity exercises (e.g., grasp release), and teaching of ADLs.. It was a 6 week's intervention in which patients got treatment protocol for 30 mints 5 times a week.
  Arms: GROUP 2

SUMMARY:
This study aims to fill this gap by investigating the effects of scapular and upper limb proprioceptive neuromuscular facilitation techniques on shoulder pain, upper limb function & gait in stroke with scapular dyskinesia. This study is a randomized control trial that includes 44 patients which were randomly divided into two groups each containing 22 participants. Experimental group will receive scapular PNF coupled with upper limb PNF and conventional physiotherapy treatment and Control group will receive only Conventional treatment.

DETAILED DESCRIPTION:
Stroke is one of the major causes of disability, cognitive decline, and mortality worldwide. This condition is recognized as the second leading cause of disability and the third leading cause of death. Scapular dyskinesia (SD) refers to the abnormal movement and function of scapula .Changes in scapular kinematics can result from altered scapular recruitment patterns , muscles performance issues and flexibility deficits in the surrounding soft tissues which may restrict normal scapular movements during daily activities.

Physical therapy is crucial for rehabilitating scapular disorders. The goal of therapeutic intervention is to restore the normal position, movement, and strength of the scapula. Specific exercises are designed to target the scapular stabilizing muscles. Proprioceptive Neuromuscular Facilitation (PNF) is a neurological technique used in therapeutic exercise that integrates functionally based diagonal movement patterns with neuromuscular facilitation techniques. This approach aims to elicit motor responses and enhance neuromuscular control and performance. This study aims to fill this gap by investigating the effects of scapular and upper limb proprioceptive neuromuscular facilitation techniques on shoulder pain, upper limb function & gait in stroke with scapular dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* • Sub-acute

  * MCA
  * Age bracket 40-65 years.
  * Gender Male or Female.
  * Gait baseline score (DGI less than 19)
  * Patients with spasticity between grades (+1 and 1) on the Modified Ashworth Scale (MAS).

Exclusion Criteria:

* • Inability to communicate/understand instructions.

  * Stroke with other neurological conditions.
  * Patient with any other psychological and medical condition.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of Upper Extremity (FMA-UE) | 6 weeks
  After a stroke, the FMA-UE is frequently used to evaluate and track recovery in hemiplegic patients.. It is a specific tool for quantifying upper limb impairment and rehabilitation outcomes in stroke patients with hemiparesis. Using a 3-point ordinal scale, the assessment rates the patient's ability to complete each task: 0 denotes incapacity to execute, 1 denotes partial completion, and 2 denotes full performance. All item scores, which range from 0 to 126, are added up to determine the final score.
Dynamic gait index (DGI) | 6 weeks
  A participant's ability to maintain walking balance while adjusting to different task demands and dynamic situations is evaluated by the Dynamic Gait Index (DGI). It is especially helpful for people who have balance and vestibular problems, as well as those who are at risk of falling. Every item has a rating between 0 and 3, where 0 denotes significant impairment and 3 denotes normal performance. 24 is the maximum possible score. A total score of less than 19 out of 24 indicates that older adults are more likely to fall, whereas a score of more than 22 indicates safe walking.
Visual Analogue Scale | 6 weeks
  Hayes and Patterson employed the visual analog scale (VAS), a pain rating tool, for the first time in 1921. A single handwritten mark is placed at one point along a 10-cm line that represents a continuum between the two ends of the scale, with "no pain" at the left end (0 cm) and the "worst pain" at the right end (10 cm). Self-identified evaluations of symptoms are used to calculate scores. The patient's discomfort is calculated by measuring the distance in centimeters between the patient's marks and the scale's beginning point (left end). The figures can be used to gauge a patient's pain progression or to compare pain across people with comparable diseases. 0 No pain, 1-3 slight pain, 4-6 moderate pain, and 7-10 excruciating pain.
10-Meter Walk Test (10MWT) | 6 weeks
  The test calculates walking speed over a brief distance in meters per second. To the closest tenth of a second, the total time spent walking six meters (m) is recorded. Then, 6 meters is divided by the whole time (in seconds) to convert this distance to m/s. The following categories apply to walking speeds: Family Ambulatory <0.40 m/s; Community Ambulator ≥0.80 m/s; Limited Community Ambulator 0.40 to <0.80 m/s

CONTACTS AND LOCATIONS:
Overall Officials: Mahat zafar, MSNMPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - HBS Hospital islamabad, Islamabad, Punjab Province
  - National institute of rehablitation medicine islamabad, Islamabad, Punjab Province

IPD SHARING:
Plan to Share IPD: No